CLINICAL TRIAL: NCT00151632
Title: Evaluation of the Benefit/Risk Ratio of a Reduction of Tacrolimus Dose in Association With Mycophenolate Mofetil on the Prevention of Complications in Adult Liver Transplantation
Brief Title: Reduction of Tacrolimus Dose in Association With Mycophenolate Mofetil After Liver Transplantation
Acronym: MMF-FK
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AFSSAPS 030200; PHRC/01-01 (Other: Rennes University Hospital); CIC0203/011
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Evidence of Liver Transplantation
Keywords: Immunosuppression; Liver transplantation; Acute graft rejection; Treatment combination
MeSH Terms: interventions — Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MMF+FK (Experimental): Low doses of tacrolimus in association with mycophenolate mofetil
  Interventions: Drug: Mycophenolate mofetil; Drug: Tacrolimus
- FK (Active Comparator): Full recommended doses of tacrolimus
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Mycophenolate mofetil — Mycophenolate mofetil is administered at a dose of 1,5 g x 2 / day for the 6 first weeks, then 1g x 2 / day until M12.
  Other Names: MMF; CELLCEPT
  Arms: MMF+FK
Drug: Tacrolimus — In arm 1: Tacrolimus is administered at half recommended dose: 0,040 mg/Kg x 2 , in order to maintain plasma levels between 6 and 10 ng/ml for the 6 first weeks, between 5 and 8 ng/ml from week 7 to M6 and between 4 and 6 ng/ml between M6 and M12.
  In arm 2: Tacrolimus is administered at the recommended dose: 0,075 mg/Kg x 2 , in order to maintain plasma levels between 12 and 20 ng/ml for the 6 first weeks, between 10 and 15 ng/ml from week 7 to week 12, between 8 and 12 ng/ml between M4 and M6 and between 6 and 10 ng/ml between M6 and M12.
  Other Names: FK; PROGRAF

SUMMARY:
The prevention of graft rejection after liver transplantation benefits nowadays from a variety of newly developed immunosuppressive agents. This allows more flexible and individualized immunoprophylaxis and gives an opportunity to reduce the long-term side effects (hypertension, renal failure, diabetes, etc.) of immunosuppression. The purpose of this study is to evaluate, in liver transplanted patients, if low doses of tacrolimus, given in combination with mycophenolate mofetil, can result in a lower rate of long-term side effects without increasing the rate of graft rejection.

DETAILED DESCRIPTION:
Tacrolimus and mycophenolate mofetil are currently approved immunosuppressive agents for the prevention of acute and chronic rejection in liver transplantation. Adverse effects of tacrolimus are dose-dependent and appear early after the onset of treatment. To prevent side effects, we propose to combine reduced doses of tacrolimus with another immunosuppressant, i.e. mycophenolate mofetil, administered at usual doses. This study evaluates the interest of this combination and, subsequently, the pharmacokinetics of mycophenolate mofetil in this therapeutic context. Patients undergoing liver transplantation will be randomized to tacrolimus at normal doses or to the combination of tacrolimus at half doses and mycophenolate mofetil. A corticotherapy will be associated in both groups. The safety will be evaluated on the number of graft rejections between day 1 after transplantation and week 48; the onset of complications (hypertension, renal failure, diabetes, etc.) will allow to evaluate the efficacy of both treatment schedules.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Primary liver transplantation
* Immunosuppressive treatment associating tacrolimus and steroids at low doses (< 20 mg/d)
* Written informed consent

Non-Inclusion Criteria:

* Pregnancy or ineffective contraception
* Immunosuppressive treatment
* Blood group incompatibility with the donor
* Autoimmune hepatitis
* Fulminant hepatitis
* Primary sclerosing cholangitis
* Combined transplantations
* Reduced liver
* Living donor
* Treated hypertension and/or diastolic pressure ≥ 90 mmHg and/or systolic pressure ≥ 140 mmHg,
* Acute or chronic renal failure(creatininemia ≥ 130 μmol/L) before transplantation
* Treated diabetes and/or fasting glycemia ≥ 7 mmol/L
* Treated hypercholesterolemia and/or cholesterolemia ≥ 7 mmol/L
* post-operative creatininemia ≥ 200 μmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2003-05; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Onset of acute rejection (criterion evaluating the risk) | between Day 1 and Week 48
Onset of at least one complication (hypertension, renal failure, diabetes) requiring a specific treatment (criterion evaluating the benefit) | between Week 9 and Week 48

SECONDARY OUTCOMES:
Onset of hypertension, renal failure, diabetes, hypercholesterolemia, or of a serious adverse effect of mycophenolate mofetil | between Day 1 and Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Karim Boudjema, MD, PhD, Study Director — CHU Rennes; Eric Bellissant, MD, PhD, Study Chair — CHU Rennes
Locations (8):
- France (8):
  - Service de Chirurgie Digestive - Hôpital de la Côte de Nacre, Caen
  - Service d'Hépatogastroentérologie - Hôpital Beaujon, Clichy
  - Service d'Hépatogastroentérologie - Hôpital Henri Mondor, Créteil
  - Chirurgie Générale et Digestive - Hôpital de La Croix Rousse, Lyon
  - Service d'Hépaogastroentérologie - Hôpital Saint Eloi, Montpellier
  - Service de Chirurgie Générale - Hôpital Cochin, Paris
  - Département de Chirurgie Viscérale - Hôpital Pontchaillou, Rennes
  - Centre Hépato-biliaire - Hôpital Paul Brousse, Villejuif

REFERENCES:
- [Background] Jain AB, Hamad I, Rakela J, Dodson F, Kramer D, Demetris J, McMichael J, Starzl TE, Fung JJ. A prospective randomized trial of tacrolimus and prednisone versus tacrolimus, prednisone, and mycophenolate mofetil in primary adult liver transplant recipients: an interim report. Transplantation. 1998 Nov 27;66(10):1395-8. doi: 10.1097/00007890-199811270-00024. PMID 9846530
- [Background] Klupp J, Glanemann M, Bechstein WO, Platz KP, Langrehr JM, Keck H, Settmacher U, Radtke C, Neuhaus R, Neuhaus P. Mycophenolate mofetil in combination with tacrolimus versus Neoral after liver transplantation. Transplant Proc. 1999 Feb-Mar;31(1-2):1113-4. doi: 10.1016/s0041-1345(98)01925-3. No abstract available. PMID 10083497